CLINICAL TRIAL: NCT05586451
Title: Muscle Activation With Acute Bouts of Blood Flow Restricted Resistance Exercise Compared to High Load Resistance Exercise in Trained Versus Untrained Adults
Brief Title: Muscle Activation With Acute Bouts of Blood Flow Restricted Resistance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University and A&M College (Other)
Responsible Party: Principal Investigator, Brian Irving, Associate Professor, Louisiana State University and A&M College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRBAM-22-0600
Record Dates: First submitted 2022-08-01; First posted 2022-10-19 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Muscle; Acute Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance Trained (Other): Resistance-trained individuals are considered those who report performing structured moderate to intense resistance exercise for at least three days per week for at least 2 years prior to study start.
  Interventions: Behavioral: Traditional High Load Resistance Exercise (HLRE); Behavioral: Low Load Resistance Exercise with Blood Flow Restriction (LLBFR); Behavioral: Moderate Load Resistance Exercise with Blood Flow Restriction (MLBFR)
- Untrained (Other): Untrained individuals are considered those that report less than two days per week of structured (> 30 minutes) moderate to vigorous-intensity aerobic exercise and less than two days per week of structured resistance training for the 3 months prior to study start.
  Interventions: Behavioral: Traditional High Load Resistance Exercise (HLRE); Behavioral: Low Load Resistance Exercise with Blood Flow Restriction (LLBFR); Behavioral: Moderate Load Resistance Exercise with Blood Flow Restriction (MLBFR)

INTERVENTIONS:
Behavioral: Traditional High Load Resistance Exercise (HLRE) — Participants will then perform 75% of tested 1RM for 3 sets of 12 repetitions at a pace of 1 repetition every 2 seconds on the dominant leg with one-minute rest between sets. After completing the HLRE protocol, participants will perform 2 post-exercise maximal voluntary contractions.
Behavioral: Low Load Resistance Exercise with Blood Flow Restriction (LLBFR) — Participants will then perform 25% of tested 1RM for sets of 30, 15, 15, and 15 repetitions on the dominant leg at a pace of 1 repetition every 2 seconds with one-minute rest between sets. Participants will be fitted with an occlusion cuff on the proximal portion of the thigh. The limb occlusion pressure will be set at 60% blood flow occlusion and remain occluded throughout the exercise (Delfi Medical Innovations Personal Tourniquet System).
Behavioral: Moderate Load Resistance Exercise with Blood Flow Restriction (MLBFR) — Participants will then perform 50% of tested 1RM for sets of 15, 8, 7, and 7 repetitions on the dominant leg at a pace of 1 repetition every 2 seconds with one-minute rest between sets. Participants will be fitted with an occlusion cuff on the proximal portion of the thigh. The limb occlusion pressure will be set at 60% blood flow occlusion and remain occluded throughout the exercise (Delfi Medical Innovations Personal Tourniquet System).

SUMMARY:
Blood flow restricted (BFR) resistance exercise has been shown to improve skeletal muscle adaptations to low load resistance exercise. One of many adaptations with resistance training is neural adaptations that occur within the first few weeks of resistance training. It has been hypothesized that these neural adaptations are blunted when using blood flow restricted exercise. Therefore, the investigators propose to examine the muscle activation created by resistance exercise with different intensities with blood flow restriction and without blood flow restriction in sedentary compared to resistance-trained individuals. The investigators will recruit and completely study up to 30, previously untrained and resistance-trained, healthy, college-aged (18-40 years) males. Participants will come in the laboratory for 5 total visits. These visits will consist of a screening/familiarization visit, a strength testing visit, and 3 acute exercise visits. The acute exercise visits will consist of 2 blood flow restricted resistance sessions at different intensities and a traditional high load resistance exercise session. The 3 acute exercise visits will be randomized. The investigators will measure muscle mass (appendicular lean mass) using Dual Energy X-Ray Absorptiometry, muscle strength and endurance using isotonic and isokinetic testing, and muscle activation using surface electromyography. The investigators will also use near infrared spectroscopy (NIRS) to measure the muscle tissue (oxygen) saturation index (TSI) in the vastus lateralis during exercise. Finally, the investigators will also draw blood before and after each exercise session to measure hormones, metabolites, and markers of inflammation using commercially available assays (e.g., ELISAs).

ELIGIBILITY:
Inclusion Criteria:

1. Capable and willing to give written informed consent
2. Capable of understanding inclusion and exclusion criteria
3. 18-40 years of age
4. A waist circumference < 40 inches.
5. No medical condition that would limit their participation in supervised exercise sessions based on the Physical Activity Readiness Questionnaire for Everyone (PARQ+)
6. No current prescription medications
7. Willing to allow researchers to use data and images (e.g., Dual Energy X-Ray Absorptiometry) for research purposes after study participation is completed
8. Either untrained or resistance-trained by the following definitions: Untrained individuals are considered those that report less than two days per week of structured (> 30 minutes) moderate to vigorous-intensity aerobic exercise and less than two days per week of structured resistance training for the 3 months prior to study start. Resistance-trained individuals are considered those who report performing structured moderate to intense resistance exercise for at least three days per week for at least 2 years prior to study start.

Exclusion Criteria:

1. Self-report history of diabetes mellitus
2. Self-report history of cardiovascular, peripheral vascular, cerebral vascular, pulmonary, or renal disease
3. Self-report or evidence of uncontrolled hypertension > 150/85 (or measured)
4. Self-report history of blood clotting disorders
5. Self-report history of deep vein thrombosis or pulmonary embolism
6. Self-report history of sickle cell trait
7. Self-report history of varicose veins
8. Self-report history of a myopathy leading to muscle loss, weakness, severe cramps or myalgia
9. Self-report history of orthopedic limitations that would preclude them from participation in a dynamic exercise program
10. Self-report history of musculoskeletal disorders (e.g., severe osteoarthritis, rheumatoid arthritis, avascular necrosis or osteonecrosis)
11. Self-report history of neurological disorders (e.g., peripheral neuropathy, amyotrophic lateral sclerosis, multiple sclerosis, fibromyalgia, Parkinson's disease)
12. Weight loss of > 10% in the last 3 months prior to screening
13. Active tobacco use including smoking, vaping, or smokeless tobacco use
14. Current consumption of > 14 alcoholic drinks per week based on self-report
15. Any other condition that, in the judgement of the Principal Investigator and/or the Medical Director of this protocol, may interfere with study participation and adherence to the protocol

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Muscle Activation Measured During Traditional High Load Resistance Exercise (HLRE) | Measurement will occur during the acute bout HLRE, which will occur during the HLRE study visit.
  Muscle (vastus lateralis) activation will be measured using surface EMG, during the knee extension exercises conducted during the acute HLRE bout.
Low Load Resistance Exercise with Blood Flow Restriction (LLBFR) | Measurement will occur during the acute bout LLBFR, which will occur during the LLBFR study visit.
  Muscle (vastus lateralis) activation will be measured using surface EMG, during the knee extension exercises conducted during the acute LLBFR bout.
Moderate Load Resistance Exercise with Blood Flow Restriction (MLBFR) | Measurement will occur during the acute bout MLBFR, which will occur during the MLBFR study visit.
  Muscle activation (vastus lateralis) will be measured using surface EMG, during the knee extension exercises conducted during the acute MLBFR bout.

SECONDARY OUTCOMES:
Change in Maximal Voluntary Contraction following HLRE | Measurements will be conducted before and immediately following the completion of the HLRE bout.
  Maximal Voluntary (isometric) Contractions will be measured using an isokinetic dynamometer before and after the acute HLRE session.
Change in Maximal Voluntary Contraction following LLBFR | Measurements will be conducted before and immediately following the completion of the LLBFR bout.
  Maximal Voluntary (isometric) Contractions will be measured using an isokinetic dynamometer before and after the acute LLBFR session.
Change in Maximal Voluntary Contraction following MLBFR | Measurements will be conducted before and immediately following the completion of the MLBFR bout.
  Maximal Voluntary (isometric) Contractions will be measured using an isokinetic dynamometer before and after the acute MLBFR session.

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Irving, Principal Investigator — School of Kinesiology
Locations (1):
- Lousiana State University, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Available upon request.